CLINICAL TRIAL: NCT04031378
Title: Phase II Randomized Study to Ablate Oligometastatic Prostate Cancer by Single Dose Radiotherapy (SDRT) With or Without Adjuvant Systemic Therapy and to Characterize Its Molecular Phenotype
Brief Title: Single Dose Radiotherapy (SDRT) With or Without Adjuvant Systemic Therapy for Oligometastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Carlo Greco, MD, M.D., Fundacao Champalimaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRELUDE
Record Dates: First submitted 2017-01-16; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Prostate Cancer; Prostate Adenocarcinoma
Keywords: Single Dose Radiotherapy; Systemic Therapy; IGRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Single Dose Radiotherapy (24 Gy) to all detectable lesions, followed by observation using PET/CT imaging studies every 6 months
  Interventions: Radiation: Single Dose Radiotherapy (24 Gy) to all detectable lesions, followed by observation
- B (Experimental): Single Dose Radiotherapy (24 Gy) to all detectable lesions followed by adjuvant systemic therapy for 6 months stratified by whether disease is castrate-sensitive (mCS-PCa) or castrate-resistant (mCR-PCa)
  Interventions: Drug: Single Dose Radiotherapy (24 Gy) to all detectable lesions followed by adjuvant systemic therapy for 6 months

INTERVENTIONS:
Radiation: Single Dose Radiotherapy (24 Gy) to all detectable lesions, followed by observation — SBRT to a single dose of 24 Gy to up to 3 sites
  Arms: A
Drug: Single Dose Radiotherapy (24 Gy) to all detectable lesions followed by adjuvant systemic therapy for 6 months — SBRT 24 Gy to up to 3 nsites, followed by by systemic therapy based on phenotype.
  Arms: B

SUMMARY:
The present study aims to optimize the use of systemic therapy relative to local tumor ablation in a prospective randomized clinical trial and to validate the existence and characterize the clinical and pathology phenotype of oligometastatic (OM) prostate cancer (OM-PCa).

For local tumor ablation we propose to use the novel non-invasive and highly effective technique of Image-Guided Single Dose Radiotherapy (SDRT), which we showed is capable of conferring long-term local relapse-free rates in ≥ 90% of metastatic PCa lesions. Concomitantly, we will develop, validate and implement a diagnostic algorithm for OM-PCa and functionally characterize Prostate Cancer Stem Cells (pCSCs) from human samples to correlate their molecular phenotypes with tumor response to treatment. The long-term aim is to define the indications, standardization of treatment protocols and outcome for OM-PCa. Response assessment will be via local control, metastasis-free survival and overall survival rates. Cases displaying the clinical OM phenotype, as disclosed via long-term disease remission following tumor ablation, will represent the basis to identify the molecular signatures of OM-PCa. These signatures will be used to develop and validate an algorithm to predict the OM phenotype upfront and define the treatment strategy that may lead to cure.

DETAILED DESCRIPTION:
Since a systemic therapy alone is incapable of permanently ablating metastatic prostate cancer (mPCa) lesions, we have designed this clinical trial to explore whether its combination with radiation ablation of low volume (≤3 detectable lesions) mPCa, using the novel and highly effective single dose radiotherapy (SDRT), will render cure of a subset of currently incurable mPCa, as achievable in other tumors at the so-called oligometastatic (OM) phase of tumor progression. Whether OM-PCa does, in fact, exist and whether it can be cured has never been systematically researched. The recent introduction of advanced diagnostic and therapeutic platforms provide new tools to address the OM paradigm in mPCa. For example, while the identification mPCa lesions is still challenging, 18F-Choline and 68Ga-Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography with Computed Tomography (PET/CT) are emerging as effective modalities for the identification of low volume metastases with a pooled sensitivity and specificity exceeding 85%. Hence, the focus of this project is to use modern diagnostic and therapeutic approaches to detect and ablate low tumor-load mPCa lesions, hypothesizing that a subset these tumors will be detected and treated at the OM phase, and may be cured. We propose that systematic studies of each tumor phenotype and their correlation with clinical outcomes will yield not only a validation of the existence of OM-PCa, but will also enable the generation of an algorithm that predicts the OM phenotype upfront and optimizes the treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate by biopsy confirmed by internal review;
* 68Ga-PSMA or 18F-Choline PET/CT evidence of limited non-visceral (1-3 detectable foci) M1a-b metastases
* All detectable lesions must be considered amenable for SDRT
* Life expectancy > 12 months
* EGOG Performance Status 0-1
* Normal bone marrow functions as defined below: Hemoglobin ≥ 9 g/dl; Absolute Neutrophil count (ANC) ≥1500/ μl; Platelets ≥ 100,000 / μl
* Signed study specific informed consent form

Exclusion Criteria:

* Overt polymetastatic disease (≥ 4 lesions or any visceral lesion) as shown by 68Ga-PSMA or 18F-Choline PET/CT
* Previous radiation therapy for OM deposits
* ECOG Performance status ≥2
* Severe, active co-morbidity
* Significant psychiatric illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-treatment abnormal laboratory values (PSA relapse) | Participants should be followed continuously, for the duration of 5 years
  Comparison of freedom from biochemical relaps over a 5 year time frame

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, M.D., Principal Investigator — Champalimaud Foundation
Locations (1):
- Fundacao Champalimaud, Lisbon, Portugal